CLINICAL TRIAL: NCT03138200
Title: The Role of Central Venous Oxygen Saturation (ScvO2) as an Indicator of Blood Transfusion in the Critically Ill
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Collaborators: Medical Centre Hungarian Defence Forces (Unknown)
Responsible Party: Principal Investigator, Zsolt Molnár, MD, PhD, DEAA, Principal Investigator, Szeged University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ScvO2 transfusion
Record Dates: First submitted 2017-03-08; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Blood Transfusion; Hemoglobinemia; Hypoxia; Anemia
Keywords: Transfusion; ScvO2; Hemoglobin
MeSH Terms: conditions — Hypoxia; Anemia | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood transfusion based on central venous oxygen saturation (Other)
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — Blood transfusion is a safe, routine procedure in which blood is given to a patient through an intravenous cannula inserted into one of the patient's veins.

SUMMARY:
Transfusion of red blood cells is an everyday practice in critical care with the primary aim of restoring adequate tissue oxygenation. However, blood transfusion may also be harmful and costly, therefore a so called restrictive transfusion regime has been suggested by recent guidelines. These transfusion guidelines consider certain levels of hemoglobin as transfusion trigger, which on its own gives little information if any about the balance between oxygen delivery (DO2) and consumption (VO2). Hence, there is a clear need for additional physiologic transfusion trigger values. One of the potentially useful and easily obtainable physiological parameters is the central venous oxygen saturation (ScvO2), which has been shown to be a potential transfusion trigger value in hemodynamically stable but anemic patients. However, the role of ScvO2 as a transfusion trigger value was examined only in a retrospective observational study and in animal experiment.

The normal value of ScvO2 in a resting adult at rest is around 70-75%, which is the product of the VO2 and DO2 relationship. Low ScvO2 usually indicates inadequate DO2. It was found in an observational study that if ScvO2>70% before transfusion due to transfusion only the value of hemoglobin increased but the value of ScvO2 did not change. This finding indicates that the DO2 may have been adequate in spite of the low hemoglobin value and the transfusion may have been unnecessary. In one of their recent animal experiments, the investigators reported that in an isovolemic-anemia model the value of ScvO2<70% was only reached when the value of hemoglobin was far less, 59 g/L, than the recommended lowest value of 70g/L as transfusion trigger by guidelines.

Despite the pathophysiological rationale and the encouraging results of retrospective studies and animal experiments, prospective randomized trials in order to test the effects of an ScvO2-assisted transfusion protocol are yet to be performed.

The aim of this study is to investigate the effects of an ScvO2-assisted transfusion protocol as compared to the guideline-based, hemoglobin levels guided transfusion practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 y)
2. Critically ill anemic but hemodynamically stable patients treated on the ICU in whom transfusion is considered by the attending physician
3. Routine ICU monitoring: invasive blood pressure, CVC, hourly urine output
4. Anemia is defined as Hb<100 g/L
5. Hemodynamic stability is defined as:

   1. heart rate (HR)<100/min,
   2. mean arterial pressure (MAP)>60 mmHg
   3. no or "minimal" requirement of noradrenaline (NA): compensation for sedation not exceeding 5 µg/min
   4. stable homeostasis:

   i. pH: 7.30-7.45 ii. HCO3 > 20 mmol/L iii. lactate < 2 mmol/L e. normal hourly urine output for the last 2 hours not facilitated by diuretics: >0.5ml/kg/h
6. Central venous catheter in situ (position in the v. cava superior confirmed by chest x-ray)

Exclusion Criteria:

1. Pregnancy
2. Head injury requiring ICP monitoring guided control of ICP
3. Shock of any origin
4. Patients with heart failure
5. Patients with renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of number of transfuion events in the two groups | 2 years
  Comparison of how many tranfusions were performed based on ScvO2 to conventional, hemoglobin based transfusion.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye
  - Department of Anaesthesia and Intensive Care, Medical Centre, Hungarian Defence Force, Budapest

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blood Observational Study Investigators of ANZICS-Clinical Trials Group; Westbrook A, Pettila V, Nichol A, Bailey MJ, Syres G, Murray L, Bellomo R, Wood E, Phillips LE, Street A, French C, Orford N, Santamaria J, Cooper DJ. Transfusion practice and guidelines in Australian and New Zealand intensive care units. Intensive Care Med. 2010 Jul;36(7):1138-46. doi: 10.1007/s00134-010-1867-8. Epub 2010 May 4. PMID 20440603
- [Background] Vallet B, Robin E, Lebuffe G. Venous oxygen saturation as a physiologic transfusion trigger. Crit Care. 2010;14(2):213. doi: 10.1186/cc8854. Epub 2010 Mar 9. PMID 20236457
- [Background] Adamczyk S, Robin E, Barreau O, Fleyfel M, Tavernier B, Lebuffe G, Vallet B. [Contribution of central venous oxygen saturation in postoperative blood transfusion decision]. Ann Fr Anesth Reanim. 2009 Jun;28(6):522-30. doi: 10.1016/j.annfar.2009.03.013. Epub 2009 May 20. French. PMID 19467825
- [Background] Kocsi S, Demeter G, Fogas J, Erces D, Kaszaki J, Molnar Z. Central venous oxygen saturation is a good indicator of altered oxygen balance in isovolemic anemia. Acta Anaesthesiol Scand. 2012 Mar;56(3):291-7. doi: 10.1111/j.1399-6576.2011.02622.x. Epub 2012 Jan 19. PMID 22260228